CLINICAL TRIAL: NCT02070757
Title: A Prospective, Randomized, Double-Blind, Multicenter, Phase 3 Study to Assess the Safety and Efficacy of Intravenous Ceftolozane/Tazobactam Compared With Meropenem in Adult Patients With Ventilated Nosocomial Pneumonia
Brief Title: Safety and Efficacy Study of Ceftolozane/Tazobactam to Treat Ventilated Nosocomial Pneumonia (MK-7625A-008)
Acronym: ASPECT-NP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625A-008; CXA-NP-11-04 (Other: Cubist Protocol Number); 163338 (Registry Identifier: JAPIC-CTI); MK-7625A-008 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Healthcare-Associated Pneumonia; Ventilator-Associated Pneumonia; Lung Diseases
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Lung Diseases | interventions — ceftolozane, tazobactam drug combination; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceftolozane/tazobactam (Experimental): Participants receive 3000 mg ceftolozane/tazobactam intravenous IV (comprising 2000 mg ceftolozane and 1000 mg tazobactam) every 8 hours for 8-14 days.
  Interventions: Drug: Ceftolozane/tazobactam
- Meropenem (Active Comparator): Participants receive 1000 mg meropenem IV every 8 hours for 8-14 days.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — Ceftolozane/tazobactam is an antibacterial consisting of a co-formulation of ceftolozane, a novel antipseudomonal cephalosporin and tazobactam, a well-established beta (β)-lactamase inhibitor (BLI) being developed for the treatment of serious bacterial infections.
  Arms: Ceftolozane/tazobactam
Drug: Meropenem — Meropenem is a broad spectrum injectable antibiotic widely used to treat serious infections such as ventilator-associated bacterial pneumonia and hospital-acquired bacterial pneumonia.
  Other Names: MERREM® IV
  Arms: Meropenem

SUMMARY:
This is a phase 3, multicenter, prospective, randomized study of intravenous (IV) ceftolozane/tazobactam versus IV meropenem in the treatment of adult participants with either ventilator-associated bacterial pneumonia (VABP) or ventilated hospital-acquired bacterial pneumonia (HABP). The primary objective is to demonstrate the non-inferiority of ceftolozane/tazobactam versus meropenem in adult participants with ventilated nosocomial pneumonia (VNP) based on the difference in Day 28 all-cause mortality rates in the Intent-to-treat (ITT) population using a non-inferiority margin of 10%.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult participants diagnosed with either VABP or ventilated HABP requiring IV antibiotic therapy;
* Intubated and on mechanical ventilation at the time of randomization;
* New or progressive infiltrate on chest radiography consistent with pneumonia;
* Presence of clinical criteria consistent with a diagnosis of ventilated nosocomial pneumonia.

Key Exclusion Criteria:

* History of moderate or severe hypersensitivity reactions to beta-lactam antibiotics;
* Prior non-study antibiotics for > 24 hours;
* Gram stain of lower respiratory tract specimen showing only gram positive bacteria;
* Active immunosuppression;
* End-stage renal disease or requirement for dialysis;
* Expected survival < 72 hours;
* Severe confounding respiratory condition (i.e., chest trauma with paradoxical respiration);
* Known or suspected community-acquired bacterial pneumonia.
* Anticipated concomitant use of any of the following medications during the course of study therapy: valproic acid or divalproex sodium. Anticipated concomitant use of serotonin re-uptake inhibitors, tricyclic antidepressants, or serotonin 5-HT1 receptor agonists (triptans), meperidine, or buspirone during the course of linezolid treatment.
* Receipt of a monoamine oxidase inhibitor within 14 days prior to the first dose of study drug or anticipated concomitant use during the course of linezolid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Xiao AJ, Miller BW, Huntington JA, Nicolau DP. Ceftolozane/tazobactam pharmacokinetic/pharmacodynamic-derived dose justification for phase 3 studies in patients with nosocomial pneumonia. J Clin Pharmacol. 2016 Jan;56(1):56-66. doi: 10.1002/jcph.566. Epub 2015 Aug 25. PMID 26096377
- [Derived] Martin-Loeches I, Shorr AF, Wunderink RG, Kollef MH, Timsit JF, Yu B, Huntington JA, Jensen E, Bruno CJ. Outcomes in participants with ventilated nosocomial pneumonia and organ failure treated with ceftolozane/tazobactam versus meropenem: a subset analysis of the phase 3, randomized, controlled ASPECT-NP trial. Ann Intensive Care. 2023 Feb 11;13(1):8. doi: 10.1186/s13613-022-01084-8. PMID 36773112
- [Derived] Kollef MH, Timsit JF, Martin-Loeches I, Wunderink RG, Huntington JA, Jensen EH, Yu B, Bruno CJ. Outcomes in participants with failure of initial antibacterial therapy for hospital-acquired/ventilator-associated bacterial pneumonia prior to enrollment in the randomized, controlled phase 3 ASPECT-NP trial of ceftolozane/tazobactam versus meropenem. Crit Care. 2022 Dec 1;26(1):373. doi: 10.1186/s13054-022-04192-w. PMID 36457059
- [Derived] Paterson DL, Bassetti M, Motyl M, Johnson MG, Castanheira M, Jensen EH, Huntington JA, Yu B, Wolf DJ, Bruno CJ. Ceftolozane/tazobactam for hospital-acquired/ventilator-associated bacterial pneumonia due to ESBL-producing Enterobacterales: a subgroup analysis of the ASPECT-NP clinical trial. J Antimicrob Chemother. 2022 Aug 25;77(9):2522-2531. doi: 10.1093/jac/dkac184. PMID 35781341
- [Derived] Shorr AF, Bruno CJ, Zhang Z, Jensen E, Gao W, Feng HP, Huntington JA, Yu B, Rhee EG, De Anda C, Basu S, Kollef MH. Ceftolozane/tazobactam probability of target attainment and outcomes in participants with augmented renal clearance from the randomized phase 3 ASPECT-NP trial. Crit Care. 2021 Oct 2;25(1):354. doi: 10.1186/s13054-021-03773-5. PMID 34600585
- [Derived] Timsit JF, Huntington JA, Wunderink RG, Shime N, Kollef MH, Kivistik U, Novacek M, Rea-Neto A, Martin-Loeches I, Yu B, Jensen EH, Butterton JR, Wolf DJ, Rhee EG, Bruno CJ. Ceftolozane/tazobactam versus meropenem in patients with ventilated hospital-acquired bacterial pneumonia: subset analysis of the ASPECT-NP randomized, controlled phase 3 trial. Crit Care. 2021 Aug 11;25(1):290. doi: 10.1186/s13054-021-03694-3. PMID 34380538
- [Derived] Castanheira M, Johnson MG, Yu B, Huntington JA, Carmelitano P, Bruno C, Rhee EG, Motyl M. Molecular Characterization of Baseline Enterobacterales and Pseudomonas aeruginosa Isolates from a Phase 3 Nosocomial Pneumonia (ASPECT-NP) Clinical Trial. Antimicrob Agents Chemother. 2021 Feb 17;65(3):e02461-20. doi: 10.1128/AAC.02461-20. Print 2021 Feb 17. PMID 33318005
- [Derived] Lodise T, Yang J, Puzniak LA, Dillon R, Kollef M. Healthcare Resource Utilization of Ceftolozane/Tazobactam Versus Meropenem for Ventilated Nosocomial Pneumonia from the Randomized, Controlled, Double-Blind ASPECT-NP Trial. Infect Dis Ther. 2020 Dec;9(4):953-966. doi: 10.1007/s40121-020-00343-0. Epub 2020 Sep 30. PMID 32996064
- [Derived] Huntington JA, Yu B, Li L, Jensen E, Bruno C, Boakye M, Zhang Z, Gao W, Feng HP, Rhee E. Outcomes in Participants with Renal Impairment from a Phase 3 Clinical Trial for Ceftolozane/Tazobactam Treatment of Nosocomial Pneumonia (ASPECT-NP). Antimicrob Agents Chemother. 2020 Nov 17;64(12):e00731-20. doi: 10.1128/AAC.00731-20. Print 2020 Nov 17. PMID 32988827
- [Derived] Kollef MH, Novacek M, Kivistik U, Rea-Neto A, Shime N, Martin-Loeches I, Timsit JF, Wunderink RG, Bruno CJ, Huntington JA, Lin G, Yu B, Butterton JR, Rhee EG. Ceftolozane-tazobactam versus meropenem for treatment of nosocomial pneumonia (ASPECT-NP): a randomised, controlled, double-blind, phase 3, non-inferiority trial. Lancet Infect Dis. 2019 Dec;19(12):1299-1311. doi: 10.1016/S1473-3099(19)30403-7. Epub 2019 Sep 25. PMID 31563344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 263 sites were opened for enrollment with the majority of participants recruited from sites in eastern Europe.
Pre-assignment Details: Randomization was stratified by diagnosis (ventilator-associated bacterial pneumonia [VABP] or ventilated hospital-acquired bacterial pneumonia [HABP]) and by age (<65 or ≥65 years). All participants randomized were included in the intent-to-treat (ITT) population.
Groups:
- Ceftolozane/Tazobactam: Participants receive 3000 mg ceftolozane/tazobactam (comprising 2000 mg ceftolozane and 1000 mg tazobactam) administered as an IV infusion every 8 hours (q8h).
- Meropenem: Participants receive 1000 mg meropenem administered as an IV infusion q8h.
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Started | 362 | 364
Treated Participants | 361 | 359
Completed | 245 | 250
Not Completed | 117 | 114
Not completed — Adverse Event | 107 | 99
Not completed — Lost to Follow-up | 7 | 4
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Investigator Decision | 0 | 2
Not completed — Discharged from Study Hospital | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam | Meropenem | Total
Number analyzed (Participants) | 362 | 364 | 726
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (16.7) | 59.5 (17.2) | 60.0 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 109 | 209
  Male | 262 | 255 | 517
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 27 | 23 | 50
  Black or African American | 10 | 4 | 14
  White | 301 | 300 | 601
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 1
  American Indian Or Alaska Native | 0 | 1 | 1
  Other | 4 | 7 | 11
  Not Reported | 19 | 27 | 46
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All Cause Mortality in the Intent-to-Treat (ITT) Population - Day 28
Description: To demonstrate the non-inferiority of ceftolozane/tazobactam versus meropenem in stratified adult participants with ventilated nosocomial pneumonia (VNP) (participants with either ventilator-associated bacterial pneumonia [VABP] or ventilated hospital-acquired bacterial pneumonia [HABP]) based on the difference in all-cause mortality rates in the intent to treat (ITT) population using a non-inferiority margin of 10%. The estimated adjusted percentage was a weighted average across all strata, constructed using Mehrotra-Railkar continuity-corrected minimum risk (MRc) stratum weights.
Time Frame: Day 28
Population: The ITT population consisted of all randomized participants with documented informed consent, regardless of whether or not they received study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 362 | 364
Percentage of Participants | 24.0 [18.83 to 27.39] | 25.3 [19.96 to 28.41]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Test type: Non-Inferiority — Meropenem minus ceftolozane/tazobactam. For ceftolozane/tazobactam to be non-inferior to meropenem the lower bound of a 2-sided 95% confidence interval (CI) for the difference between treatment groups had to be ≥ -10%; Difference in Percentage of Participants = 1.1, 95% CI 2-sided [-5.13 to 7.39] — The % difference between groups is the weighted proportion difference using MRc stratum weights for diagnosis and age categories. The 95% CI was stratified Wilson intervals for group percentages and a stratified Newcombe interval for the difference

2. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at the Test-of-Cure (TOC) Visit in the Intent-to-Treat (ITT) Population
Description: To demonstrate the non-inferiority of ceftolozane/tazobactam versus meropenem in adult participants with ventilated nosocomial pneumonia (VNP) at the TOC visit (7 to 14 days after the end-of-therapy [EOT] visit) using a non-inferiority margin of 12.5%. Clinical response at the TOC visit was defined as cure (complete resolution with no new signs of VNP), failure (progression, relapse or recurrence of VNP) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate unless the clinical outcome at the EOT visit was failure. The estimated adjusted percentage was a weighted average across all strata, constructed using Mehrotra-Railkar continuity-corrected minimum risk (MRc) stratum weights.
Time Frame: 7 to 14 days after last dose of study drug (Up to ~Day 30)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 362 | 364
Percentage of Participants | 54.4 [49.47 to 59.60] | 53.3 [48.44 to 58.54]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Test type: Non-Inferiority — Clinical Response difference is calculated as ceftolozane/tazobactam minus meropenem. For ceftolozane/tazobactam to be non-inferior to meropenem the lower bound of a 2-sided 95% confidence interval (CI) for the difference between treatment groups had to be ≥ -12.5%; Difference in percentage of participants = 1.1, 95% CI 2-sided [-6.17 to 8.29] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With All Cause Mortality in the Microbiological Intent-to-Treat (mITT) Population - Day 28
Description: To compare the all cause mortality rates of participants in the ceftolozane/tazobactam versus meropenem arms in microbiological intent-to-treat (mITT) population.
Time Frame: Day 28
Population: The mITT population was a subset of the ITT population that included any participant who received any amount of study drug and had at least 1 bacterial respiratory pathogen isolated from the baseline LRT culture that was susceptible to at least 1 of the study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 264 | 247
Percentage of Participants | 20.1 [15.12 to 24.50] | 25.5 [18.89 to 29.35]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — The % difference is the weighted proportion difference using Mehrotra-Railkar continuity-corrected-minimum risk (MRc) stratum weights for strata of diagnosis (VABP, ventilated HABP) and age (<65, >=65) categories; Difference in Percentage of Participants = 4.4, 95% CI 2-sided [-2.83 to 11.75] — The 95% confidence interval (CI) were stratified Wilson intervals for the treatment group percentages and a stratified Newcombe interval for the treatment difference, constructed using the MRc stratum weights

4. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at the Test-of-Cure (TOC) Visit in the Clinically Evaluable (CE) Population
Description: To compare the clinical response rates of ceftolozane/tazobactam versus meropenem in adult participants with VNP (participants with either ventilator-associated bacterial pneumonia [VABP] or ventilated hospital-acquired bacterial pneumonia [HABP]) at the TOC visit in the CE population. Clinical response at the TOC visit was defined as cure (complete resolution with no new signs of VNP), failure (progression, relapse or recurrence of VNP) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate unless the clinical outcome at the EOT visit was failure. The data-as-observed (DAO) approach was used where participants with missing clinical responses, including indeterminate outcomes, are excluded from the analysis population.
Time Frame: 7 to 14 days after last dose of study drug (Up to ~Day 30)
Population: The CE population was a subset of the ITT population that included any participant who received study drug, adhered to the study protocol through the TOC visit, and had an evaluable clinical outcome (either Cure or Failure) at the TOC visit (or were classified as a clinical failure prior to the TOC visit).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 218 | 221
Percentage of Participants | 63.8 [57.50 to 70.11] | 64.7 [58.83 to 71.19]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = -1.3, 95% CI 2-sided [-10.21 to 7.67] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants With Per-Participant Microbiological Response of Cure or Presumed Cure at the Test-of-Cure (TOC) Visit in the Microbiologically Evaluable (ME) Population
Description: To compare the per-participant microbiological response rates of ceftolozane/tazobactam versus meropenem at the TOC visit in the microbiologically evaluable (ME) population. The per-participant microbiological response will be determined based on the individual microbiological outcomes for each baseline pathogen. A microbiological response at the TOC visit was defined as cure (baseline pathogens eradicated), failure (baseline pathogen is persistent) or indeterminate (no evaluable respiratory material). A favorable microbiological response is a microbiological cure or presumed cure. The data-as-observed (DAO) approach was used where participants with missing clinical responses, including indeterminate outcomes, are excluded from the analysis population.
Time Frame: 7 to 14 days after last dose of study drug (Up to ~Day 30)
Population: The ME population was a subset of the mITT population that included any participants who adhered to the study protocol through the TOC visit, had an evaluable clinical outcome (Cure or Failure) at the TOC visit and had at least 1 bacterial respiratory pathogen (at the appropriate CFU/mL threshold) isolated from the baseline LRT culture.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 115 | 118
Percentage of Participants | 70.4 [61.37 to 77.55] | 62.7 [54.12 to 71.24]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = 7.0, 95% CI [-5.11 to 18.93] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants With Microbiological Response of Eradication or Presumed Eradication, by Pathogen, at the Test-of-Cure (TOC) Visit in the Microbiologically Evaluable (ME) Population (>=10 Isolates at Baseline)
Description: To compare the percentage of participants with a microbiological outcome of eradication or presumed eradication, by pathogen. The microbiological outcome was classified as "eradication", "presumed eradication", "persistence", 'presumed persistence", "indeterminate" or "recurrence." "Eradication" was defined as a ≥1- log reduction in bacterial burden of the original baseline LRT pathogen AND a per pathogen count of ≤10^4 colony-forming unit (CFU)/mL for endotracheal aspirate (ETA) or sputum specimens, ≤10^3 CFU/mL for a bronchoalveolar lavage (BAL) specimen, or ≤10^2 CFU/mL for a protected brush specimen (PBS) from a follow-up LRT culture. Presumed eradication was defined as an absence of material to culture (e.g. inability to obtain a culture in an extubated patient) in a patient deemed a clinical cure.
Time Frame: 7 to 14 days after last dose of study drug (Up to ~Day 30)
Population: The ME population included any participants in the mITT who adhered to the protocol, had an evaluable clinical outcome at TOC and at least 1 pathogen isolated from the baseline LRT culture at the appropriate CFU/mL threshold. The number analyzed per pathogen represents the number of participants in the ME population with that specific pathogen.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 115 | 118
Percentage of Participants
  Gram-Negative: number analyzed (Participants) | 113 | 117
  Gram-Negative | 69.9 [60.91 to 77.60] | 62.4 [53.35 to 70.64]
  Pseudomonas aeruginosa: number analyzed (Participants) | 29 | 38
  Pseudomonas aeruginosa | 79.3 [61.61 to 90.15] | 55.3 [39.71 to 69.85]
  Enterobacteriaceae: number analyzed (Participants) | 83 | 90
  Enterobacteriaceae | 68.7 [58.06 to 77.64] | 65.6 [55.28 to 74.55]
  Escherichia coli: number analyzed (Participants) | 23 | 23
  Escherichia coli | 78.3 [58.10 to 90.34] | 73.9 [53.53 to 87.45]
  Klebsiella pneumoniae: number analyzed (Participants) | 42 | 48
  Klebsiella pneumoniae | 71.4 [56.43 to 82.83] | 66.7 [52.54 to 78.32]
  Proteus mirabilis: number analyzed (Participants) | 11 | 10
  Proteus mirabilis | 63.6 [35.38 to 84.83] | 70.0 [39.68 to 89.22]
  Haemophilus influenzae: number analyzed (Participants) | 12 | 8
  Haemophilus influenzae | 91.7 [64.61 to 98.51] | 50.0 [21.52 to 78.48]
  Enterobacter cloacae: number analyzed (Participants) | 7 | 8
  Enterobacter cloacae | 57.1 [25.05 to 84.18] | 75.0 [40.93 to 92.85]
  Klebsiella oxytoca: number analyzed (Participants) | 8 | 7
  Klebsiella oxytoca | 87.5 [52.91 to 97.76] | 57.1 [25.05 to 84.18]
  Serratia marcescens: number analyzed (Participants) | 5 | 6
  Serratia marcescens | 40.0 [11.76 to 76.93] | 50.0 [18.76 to 81.24]
  Acinetobacter baumannii: number analyzed (Participants) | 6 | 5
  Acinetobacter baumannii | 33.3 [9.68 to 70.00] | 80.0 [37.55 to 96.38]

7. Secondary Outcome: Percentage of Participants With All-Cause Mortality in the Intent-to-Treat (ITT) Population - Day 14
Description: To compare the all cause mortality rates of participants (ceftolozane/tazobactam versus meropenem arms). Participants whose Day 14 mortality outcomes are missing or unknown are analysed as deceased.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 362 | 364
Percentage of Participants | 14.1 [10.48 to 17.57] | 12.9 [9.31 to 15.86]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = -1.4, 95% CI 2-sided [-6.41 to 3.57] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at the End-of-Therapy (EOT) Visit in the Intent-to-Treat (ITT) Population
Description: To compare the clinical response rates at the EOT visit for ceftolozane/tazobactam versus meropenem. Clinical response at the EOT visit was defined as cure (complete resolution with no new signs of VNP), failure (progression, relapse or recurrence of VNP) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate.
Time Frame: Within 24 hours after last dose of study drug (Up to ~Day 15)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 362 | 364
Percentage of Participants | 66.0 [61.38 to 71.03] | 66.8 [62.31 to 71.77]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = -0.8, 95% CI 2-sided [-7.67 to 6.04] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Percentage of Participants With Per-Participant Microbiological Response of Cure or Presumed Cure at the End-of-Therapy (EOT) Visit in the Microbiologically Evaluable (ME) Population
Description: To compare the microbiological response rates of ceftolozane/tazobactam versus meropenem at the EOT visit. The per-participant microbiological response will be determined based on the individual microbiological outcomes for each baseline pathogen. A microbiological response at the EOT visit was defined as cure (baseline pathogens eradicated), failure (baseline pathogen is persistent) or indeterminate (no evaluable respiratory material). A favorable microbiological response is a microbiological cure or presumed cure. The data-as-observed (DAO) approach was used where participants with missing clinical responses, including indeterminate outcomes, are excluded from the analysis population.
Time Frame: Within 24 hours after last dose of study drug (Up to ~Day 15)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 264 | 247
Percentage of Participants | 80.9 [71.51 to 86.33] | 78.8 [70.25 to 84.90]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = 1.6, 95% CI 2-sided [-8.91 to 12.02] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Percentage of Participants With Clinical Response of Clinical Cure at the Late Follow-up (LFU) Visit in the Clinically Evaluable (CE) Population
Description: To compare the clinical response rates at the Late Follow-up (LFU) visit for ceftolozane/tazobactam versus meropenem in the CE population. Clinical response at the LFU visit will be classified as sustained cure, relapse, or indeterminate only in participants deemed a clinical cure at the TOC visit. A favorable clinical response is "sustained clinical cure."
Time Frame: 28 to 35 days after the last dose of study drug (Up to ~Day 50)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 218 | 221
Percentage of Participants | 52.8 [90.10 to 97.99] | 51.6 [85.86 to 95.72]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage of Participants; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage of Participants = 3.3, 95% CI 2-sided [-3.38 to 10.44] — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Percentage of Participants Who Report 1 or More Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 35 days after last dose of study drug (Up to ~Day 50)
Population: All safety analyses were based on a subset of the ITT population (the Safety Population), which included randomized participants who received any amount (i.e., full or partial dose) of study drug. All participants received their randomly assigned treatments, and no participants with important deviations were excluded from the safety population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 361 | 359
Percentage of Participants | 85.9 | 83.3

12. Secondary Outcome: Percentage of Participants With Any Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to 35 days after last dose of study drug (Up to ~Day 50)
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 361 | 359
Percentage of Participants | 42.1 | 35.9

13. Secondary Outcome: Percentage of Participants Discontinuing Study Drug Due to an Adverse Event (AE)
Description: as for outcome 11
Time Frame: Up to 14 days after the first dose of study drug (Up to ~Day 15)
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 361 | 359
Percentage of Participants | 10.2 | 11.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 35 days after last dose of study drug (Up to ~Day 50)
Description: All safety analyses were based on a subset of the ITT population who received any amount (i.e., full or partial dose) of study drug (the Safety Population). All participants received their randomly assigned treatments, and no participants with important deviations were excluded from the safety population. Discontinuations due to adverse events (AEs) include deaths.
Arm/Group | Ceftolozane/Tazobactam | Meropenem
All-Cause Mortality (participants affected / at risk) | 105/361 | 101/359
Serious Adverse Events (participants affected / at risk) | 152/361 | 129/359
Other Adverse Events (participants affected / at risk) | 113/361 | 111/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=361) | Meropenem (N=359)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 8 (9) | 6 (6)
Cardiac failure (Cardiac disorders) | 7 (7) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 9 (9) | 7 (7)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 4 (4)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 3 (3)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Brain death (General disorders) | 3 (3) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 4 (4)
Multi-organ failure (General disorders) | 14 (14) | 9 (9)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
CNS ventriculitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endotoxaemia (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 3 (3)
Peritonitis (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 3 (3)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 13 (13) | 14 (14)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Apallic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1)
Brain midline shift (Nervous system disorders) | 4 (4) | 1 (1)
Brain oedema (Nervous system disorders) | 8 (8) | 8 (8)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 5 (5) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 9 (9) | 3 (3)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 2 (2)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=361) | Meropenem (N=359)
Anaemia (Blood and lymphatic system disorders) | 32 (32) | 38 (45)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 25 (28)
Urinary tract infection (Infections and infestations) | 23 (24) | 25 (27)
Alanine aminotransferase increased (Investigations) | 20 (21) | 14 (14)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 20 (24)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 25 (30) | 17 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will review proposed publication within forty five (45) calendar days and reserves the right to defer such publication an additional forty five (45) calendar days to protect Sponsor's intellectual property as applicable. If a joint manuscript has not been submitted for publication within twelve (12) months of completion or termination of Trial at all participating sites, Principal Investigator is free to publish separately, subject to the other requirements of this Agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT02070757/Prot_SAP_000.pdf